CLINICAL TRIAL: NCT05086653
Title: The Management of Left Atrial Appendage Perforation Complicated by Cardiac Tamponade During Left Atrial Appendage Occluder Device Deployment
Brief Title: Complications From Left Atrial Appendage Occluder
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Siew Yoek Chan, general practitioner, Kaohsiung Medical University
Other Study IDs: LAA
Record Dates: First submitted 2021-09-27; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation; Cardiac Perforation; Cardiac Tamponade
MeSH Terms: conditions — Atrial Fibrillation; Cardiac Tamponade | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery — Sutured by Prolene 3-0 with two layers of pledge

SUMMARY:
The following case reported a rare complication of left atrial appendage perforation complicated by cardiac tamponade during LAAO device deployment and its corresponding surgical management

ELIGIBILITY:
Inclusion Criteria:

* 73-year-old woman with CHA2DS2-VASc score 4

Exclusion Criteria:

* nil

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: one female patient involved
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Treatment related adverse events | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Division of Cardiovascular Surgery, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
This is a case report